CLINICAL TRIAL: NCT06559306
Title: A Two-Part Multicenter, Double-Blind, Randomized Placebo-Controlled Study to Evaluate Efficacy and Safety and the Maintenance of Effect of 20-(Milligram) mg Seltorexant as Adjunctive Therapy to Antidepressants in Adult and Elderly Patients With Major Depressive Disorder With Insomnia Symptoms
Brief Title: Phase 3 Study of Adjunctive Treatment With Seltorexant in Adult and Elderly Participants With Major Depressive Disorder and Insomnia Symptoms
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42847922MDD3003; 42847922MDD3003 (Other: Janssen Research & Development, LLC); 2023-509070-36-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Seltorexant (Experimental): Participants will receive seltorexant orally once daily for 6 weeks during the double-blind (DB) treatment phase in Part 1 of the study. Participants who do not proceed to Part 2 of the study will undergo a post-treatment follow-up phase, after the DB treatment phase in Part 1 and will continue to take their single baseline selective serotonin reuptake inhibitor (SSRI)/serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant throughout the study.
  Interventions: Drug: Seltorexant; Drug: Selective Serotonin Reuptake Inhibitor (SSRI)/Serotonin-Norepinephrine Reuptake Inhibitor (SNRI)
- Part 1: Placebo (Placebo Comparator): Participants will receive matching placebo orally once daily for 6 weeks during the DB treatment phase in Part 1 of the study. Participants who do not proceed to Part 2 of the study will undergo a post-treatment follow-up phase, after the DB treatment phase in Part 1 and will continue to take their single baseline SSRI/SNRI antidepressant throughout the study.
  Interventions: Drug: Placebo; Drug: Selective Serotonin Reuptake Inhibitor (SSRI)/Serotonin-Norepinephrine Reuptake Inhibitor (SNRI)
- Part 2: Open Label (OL) Seltorexant (Experimental): All participants who complete Part 1, and who meet eligibility criteria for Part 2, as well as direct entry participants, will enter Part 2 of the study. In Part 2 open-label phases (induction and stabilization) all participants (newly enrolled direct entry participants and Part 1 roll-over participants) will receive seltorexant orally in addition to their background SSRI/SNRI treatment.
  Interventions: Drug: Seltorexant; Drug: Selective Serotonin Reuptake Inhibitor (SSRI)/Serotonin-Norepinephrine Reuptake Inhibitor (SNRI)
- Part 2: DB Seltorexant (Experimental): All participants who complete Part 1, and who meet eligibility criteria for Part 2, as well as direct entry participants, will enter Part 2 of the study. Participants who achieve a stable response during the open-label phase will receive treatment with seltorexant orally once daily during DB Maintenance Phase in Part 2 of the study. Participants will continue to take their single baseline SSRI/SNRI antidepressant throughout the study.
  Interventions: Drug: Seltorexant; Drug: Selective Serotonin Reuptake Inhibitor (SSRI)/Serotonin-Norepinephrine Reuptake Inhibitor (SNRI)
- Part 2: DB Placebo (Placebo Comparator): All participants who complete Part 1, and who meet eligibility criteria for Part 2, as well as direct entry participants, will enter Part 2 of the study. Participants who achieve a stable response during the open-label phases will receive treatment with matching placebo orally once daily during DB Maintenance Phase in Part 2 of the study. Participants will continue to take their single baseline SSRI/SNRI antidepressant throughout the study.
  Interventions: Drug: Placebo; Drug: Selective Serotonin Reuptake Inhibitor (SSRI)/Serotonin-Norepinephrine Reuptake Inhibitor (SNRI)

INTERVENTIONS:
Drug: Seltorexant — Seltorexant will be administered orally.
  Other Names: JNJ 42847922
  Arms: Part 1: Seltorexant; Part 2: DB Seltorexant; Part 2: Open Label (OL) Seltorexant
Drug: Placebo — Matching Placebo tablets will be administered orally.
  Arms: Part 1: Placebo; Part 2: DB Placebo
Drug: Selective Serotonin Reuptake Inhibitor (SSRI)/Serotonin-Norepinephrine Reuptake Inhibitor (SNRI) — SSRI/SNRI will be administered orally.

SUMMARY:
The purpose of this study is to know how well seltorexant works, and also to evaluate safety and maintenance effect of seltorexant compared with placebo as an adjunctive therapy to an antidepressant in improving depressive symptoms in participants with major depressive disorder with insomnia symptoms (MDDIS) who have had an inadequate response to current antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI).

ELIGIBILITY:
Inclusion Criteria:

Participants in part 1 and direct enrollers to part 2:

* Meet DSM-5 MDD, without psychotic features based upon clinical assessment and confirmed by the structured clinical interview for DSM-5 Axis I disorders-clinical trials version (SCID-CT) diagnosed with first depressive episode prior to age 60
* Have had an inadequate response to at least 1 but no more than 2 antidepressants, administered at an adequate dose and duration in the current episode of depression. An inadequate response is defined as less than (<) 50% reduction but with some improvement (that is, improvement greater than [>] 0%) in depressive symptom severity with residual symptoms other than insomnia present, and overall good tolerability, as assessed by the MGH-ATRQ, and this must include the participant's current antidepressant treatment
* Is receiving and tolerating well any one of the following SSRI or SNRI for depressive symptoms at screening, in any formulation and available in the participating country: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at therapeutic dose level) for at least 6 weeks
* Having a major depressive episode of at least moderate severity, as assessed with 17-item Hamilton Depression Rating Scale, implemented through the Structured Interview Guide (SIGH-D) in a blinded manner at screening and must not demonstrate a clinically significant improvement from the beginning to end of screening.

Participants entering after completing part 1:

* Must have completed Part 1 DB treatment phase
* Can consistently tolerate study drug (at the end of Part 1), and there is no additional safety risk for the participant if they proceed to Part 2
* Was able to consistently follow the study procedures in Part 1 as judged by the investigator.
* Must be medically stable based on clinical laboratory tests

Exclusion Criteria:

* Has a recent (last 3 months) history of, or current signs and symptoms of, severe renal insufficiency clinically significant or unstable cardiovascular, respiratory, gastrointestinal, neurologic, hematologic, rheumatologic, immunologic or endocrine disorders and uncontrolled Type 1 or Type 2 diabetes mellitus
* Has a history of narcolepsy and seizures
* Has current signs/symptoms of hypothyroidism or hyperthyroidism
* Participants taking thyroid supplementation for antidepressant purposes
* Has Cushing's disease, Addison's disease, primary amenorrhea, or other evidence of significant medical disorders of the HPA axis

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Day 43 | Baseline, Day 43
  The MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Part 2: Time from Randomization to the First Relapse in Participants Who Achieve a Stable Response | Time from randomization to the first Relapse during the maintenance phase (up to 2 years and 10 months)
  Stable response is defined as a greater than equal to (>=) 50 percent (%) reduction in the MADRS total score for the last 3 consecutive visits of the OL stabilization Phase, as assessed by the site investigator. Time from randomization to the first relapse during the DB maintenance phase in participants who achieve a stable response at the end of OL seltorexant treatment will be reported.

SECONDARY OUTCOMES:
Part 1: Change from Baseline in the MADRS Without Sleep Item (MADRS-WOSI) Total Score at Day 43 | Baseline, Day 43
  MADRS-WOSI considered 9 of the 10 MADRS items, excluding "reduced sleep" item. The total score ranged from 0 to 54, with higher scores corresponding to greater symptom severity.
Part 1: Change from Baseline in Sleep Disturbance Using the Patient Reported Outcome Measurement Information System-Sleep Disturbance (PROMIS-SD) Short Form 8a T-score at Day 43 | Baseline, Day 43
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 8-item short form will be used in this study, in which responses are scored 1 to 5 for each item. T-score for the PROMIS-SD scales represent the value obtained after using a conversion table to convert the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. Higher overall score indicates more sleep disturbance.
Part 1: Change from Baseline in the MADRS-6 Total Score at Day 43 | Baseline, Day 43
  The MADRS-6 scale is a clinician-administered questionnaire used to measure the severity of major depressive disorder (MDD) symptoms. The MADRS-6 scale is a subset of the MADRS -10 scale, comprised of the following individual questionnaire items: apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thoughts. Scores range from 0 (no apparent symptoms) to 36 (most severe symptoms).
Part 1: Percentage of Participants with Response on Depressive Symptoms Scale Based on Montgomery-Asberg Depression Rating Scale (MADRS) Total score From Baseline to Day 43 | From Baseline to Day 43
  Responders are defined as participants with >= 50 percent improvement in the MADRS total score from baseline to Day 43.
Part 1: Change from Baseline in Sleep Disturbance Using the Patient Reported Outcome Measurement Information System-Sleep Disturbance (PROMIS-SD) Short Form (4a) T-score at Day 43 | Baseline, Day 43
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 4-item short form will be used in this study, in which responses are scored 1 to 5 for each item. T-score for the PROMIS-SD scales represent the value obtained after using a conversion table to convert the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 4-item form, the lowest possible raw score is 4; the highest possible raw score is 20. Higher overall score indicates more sleep disturbance.
Part 1: Change from Baseline in Sleep Disturbance Using the Patient Reported Outcome Measurement Information System-Sleep Disturbance (PROMIS-SD) Short Form (10a) T-score at Day 43 | Baseline, Day 43
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 10-item short form will be used, in which responses are scored 1 to 5 for each item. T-score for the PROMIS-SD scales represent the value obtained after using a conversion table to convert the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 10-item form, the lowest possible raw score is 10; the highest possible raw score is 50. Higher overall score indicates more sleep disturbance.
Part 1: Change from Baseline in Patient Health Questionnaire, 9-Item (PHQ-9) Total Score at Day 43 | Baseline, Day 43
  The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the diagnostic and statistical manual of mental disorders-5th edition (DSM-5) major depressive disorder (MDD) criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Part 2: Time from Randomization to the First Relapse in Participants Who Achieve a Stable Remission | Time from randomization to the first relapse during the maintenance phase (up to 2 years and 10 months)
  Stable remission is defined as MADRS total score less than or equal to (<=)10 and CGI-S <= 2 for at least 4 consecutive weeks of the OL stabilization Phase. Time from randomization to the first relapse during the DB maintenance phase in participants who achieve stable remission at the end of the OL seltorexant treatment will be reported.
Part 2: Change from Baseline to Endpoint of the DB Maintenance Phase in Sleep Disturbance Using the PROMIS-SD Short Form (8a) T-Score | From Baseline (Day 1 in the DB treatment maintenance Phase) until end point of the DB maintenance phase (that is up to Day 337)
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 8-item short form will be used in this study, in which responses are scored 1 to 5 for each item. T-score for the PROMIS-SD scales represent the value obtained after using a conversion table to convert the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. Higher overall score indicates more sleep disturbance.
Part 2: Change from Baseline to Endpoint of the DB Maintenance Phase in Sleep Disturbance Using the PROMIS-SD Short Form (4a) T-Score | From Baseline (Day 1 in the DB treatment maintenance Phase) until end point of the DB maintenance phase (that is up to Day 337)
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 4-item short form will be used in this study, in which responses are scored 1 to 5 for each item. T-score for the PROMIS-SD scales represent the value obtained after using a conversion table to convert the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 4-item form, the lowest possible raw score is 4; the highest possible raw score is 20. Higher overall score indicates more sleep disturbance.
Part 2: Change from Baseline in Sleep Disturbance Using the Patient Reported Outcome Measurement Information System-Sleep Disturbance (PROMIS-SD) Short Form (10a) T-score at Day 43 | Baseline, Day 43
  The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 10-item short form will be used, in which responses are scored 1 to 5 for each item. T-score for the PROMIS-SD scales represent the value obtained after using a conversion table to convert the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 10-item form, the lowest possible raw score is 10; the highest possible raw score is 50. Higher overall score indicates more sleep disturbance.
Part 2: Change from Baseline to Endpoint of the DB Maintenance Phase in MADRS Total Score | From Baseline (Day 1 in the DB treatment maintenance Phase) until end point of the DB maintenance phase (that is up to Day 337)
  The MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Part 2: Change from Baseline to Endpoint of DB Maintenance Phase in PHQ-9 Score | From Baseline (Day 1 in the DB Treatment Maintenance Phase) Until End Point of the DB Maintenance Phase (that is, up to Day 337)
  The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the DSM-5 MDD criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Change From Baseline to Endpoint of the DB Maintenance Phase in the MADRS-6 score | From Baseline (Day 1 in the DB treatment maintenance Phase) until end point of the DB maintenance phase (that is up to Day 337)
  The MADRS-6 scale is a clinician-administered questionnaire used to measure the severity of MDD symptoms. The MADRS-6 scale is a subset of the MADRS -10 scale, comprised of the following individual questionnaire items: apparent sadness, reported sadness, inner tension, lassitude, inability to feel, and pessimistic thoughts. Scores range from 0 (no apparent symptoms) to 36 (most severe symptoms).
Change from Baseline to Endpoint of the DB Maintenance Phase in the MADRS symptoms other than insomnia MADRS Without Sleep Item (MADRS-WOSI) | From Baseline (Day 1 in the DB treatment maintenance Phase) until end point of the DB maintenance phase (that is up to Day 337)
  MADRS-WOSI considered 9 of the 10 MADRS items, excluding "reduced sleep" item. The total score ranged from 0 to 54, with higher scores corresponding to greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trail, Study Director — Janssen Research & Development, LLC
Locations (196):
- United States (84):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - University of Arizona, Tucson, Arizona
  - SanRo Clinical Research Group LLC WCG Clinical Network, Bryant, Arkansas
  - Preferred Research Partners, Little Rock, Arkansas
  - PAMOJA Clinical Institute LLC, Anaheim, California
  - Axiom Research, Colton, California
  - Elite Research Network, Encino, California
  - Behavioral Research Specialists LLC, Glendale, California
  - WR PRI Los Alamitos, Los Alamitos, California
  - Excell Research Inc, Oceanside, California
  - Prospective Research Innovations Inc, Rancho Cucamonga, California
  - Anderson Clinical Research, Redlands, California
  - Lumos Clinical Research Center LLC, San Jose, California
  - Syrentis Clinical Research, Santa Ana, California
  - California Neuroscience Research, Sherman Oaks, California
  - Mountain View Clinical Research, Denver, Colorado
  - UConn Health Center, Farmington, Connecticut
  - Clinical Research of Brandon, Brandon, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Clinical NeuroScience Solutions Inc, Jacksonville, Florida
  - Multi Specialty Research Associates Inc, Lake City, Florida
  - Alcanza Clinical Research, Largo, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Nuovida Research Center, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - Nova Psychiatry INC, Orlando, Florida
  - Florida Center for TMS, Saint Augustine, Florida
  - University of South Florida, Tampa, Florida
  - Psych Me Medical Research Inc, Tampa, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Health Synergy Clinical Research, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Advanced Discovery Research, Atlanta, Georgia
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Peachford Hospital-Atlanta Behavorial Research, Dunwoody, Georgia
  - Accelerated Clinical Research Group LLC, Peachtree Corners, Georgia
  - iResearch Savannah, Savannah, Georgia
  - Renew Health Clinical Research, Snellville, Georgia
  - Northwestern University, Chicago, Illinois
  - MetroMed Clinical Research, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Revive Research Institute, Elgin, Illinois
  - Baber Research Group, Naperville, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - Adams Clinical LLC, Watertown, Massachusetts
  - Mankato Clinic, Mankato, Minnesota
  - Redbird Research, Las Vegas, Nevada
  - Oasis Clinical Research LLC, Las Vegas, Nevada
  - ActivMed Practices and Research, Portsmouth, New Hampshire
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - University at Buffalo Psychiatry, Buffalo, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Fieve Clinical Research Inc, New York, New York
  - Hapworth Psychiatric Medical PLLC, New York, New York
  - Lucian Miron Manu MD Psychiatry PC, Woodbury, New York
  - IMA Clinical Research PC, Hickory, North Carolina
  - Haidar Almhana Nieding, Avon Lake, Ohio
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas at Austin, Austin, Texas
  - BioBehavioral Research of Austin PC, Austin, Texas
  - Houston Clinical Trials LLC, Bellaire, Texas
  - Relaro Medical Trials, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - VAST Clinical Research, Garland, Texas
  - Baylor College of Medicine, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - R and H Clinical Research, Stafford, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Cedar Clinical Research, Draper, Utah
  - Core Clinical Research, Everett, Washington
- Argentina (8):
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Centro Medico Luquez, Córdoba
  - Sanatorio Prof Leon S Morra S A, Córdoba
  - INSA Instituto de Neurociencias San Agustín, La Plata
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
  - Clinica El Jardin, Santiago del Estero
- Brazil (12):
  - L2IP Instituto de Pesquisas Clinicas, Brasília
  - CAEP Centro Avancado De Estudos E Pesquisas, Campinas
  - Sociedade Literaria e Caritativa Santo Agostinho Hospital Sao Jose, Criciúma
  - Universidade Federal do Rio Grande do Norte Hospital Universitario Onofre Lopes, Natal
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Hospital De Clinicas De Porto Alegre, Porto Alegre
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia INSCER Instituto do Cerebro do Rio Grande do Sul, Porto Alegre
  - Ruschel Medicina e Pesquisa Clínica Ltda, Rio de Janeiro
  - Centro Integrado Facili, São Bernardo do Campo
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - BR Trials, São Paulo
- Bulgaria (7):
  - Mental Health Center Prof. Dr. Ivan Temkov, Burgas
  - UMHAT 'Sveti Georgi'- Plovdiv, Psychiatry Clinic, Plovdiv
  - Medical Center St. Naum, Sofia
  - Centre for Mental Health Prof.N.Shipkovenski EOOD, Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - Medical Center ZaraMed, Stara Zagora
  - Diagnostic Consulting Center Mladost - M Varna, Varna
- Czechia (6):
  - Medipa S R O, Brno
  - A Shine S R O, Pilsen
  - Clintrial s r o, Prague
  - Neuropsychiatrie Petrska sro, Prague
  - Pragtis S R O, Prague
  - Medical Services Prague S R O, Prague
- Italy (10):
  - Territorial Social Health Authority of the Spedali Civili of Brescia, Brescia
  - Azienda Ospedaliero Univ. Policlinico Gaspare Rodolico, Catania
  - Universita D Annunzio, Chieti
  - IRCCS Aor San Martino IST, Genova
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
  - Ospedale S Francesco d Assisi, Salerno
  - A O Universitaria Senese Ospedale Santa Maria alle Scotte, Siena
- Mexico (7):
  - Health Pharma Professional Research, Mexico City
  - Ketamine Mexico S de RL de C V, Mexico City
  - Gabipros SC, Mexico City
  - Instituto de Informacion e Investigacion en Salud Mental A.C., Monterrey
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
  - Centro de Estudios Clinicos y Especialidades Medicas S C, Nuevo León
  - Hospital Lomas de San Luis Internacional, San Luis de Potosi
- Poland (11):
  - Centrum Medyczne Intercor Sp z o o, Bydgoszcz
  - Osrodek Badan Klinicznych CLINSANTE S C Ewa Galczak Nowak Malgorzata Trzaska, Bydgoszcz
  - PROMENTE Sp. z o.o., Bydgoszcz
  - Centrum Zdrowia Alcea, Gdansk
  - Specjalistyczna Praktyka Lekarska Piotr Zalitacz, Gorlice
  - Przychodnie Grudziadz sp. z o.o., Grudziądz
  - Clinic BBP, Katowice
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Praktyka Lekarska dr n med Malgorzata Wojtanowska Bogacka, Poznan
  - Szpital Nowowiejski Osrodek Badan Klinicznych, Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
- Portugal (9):
  - Uls Braga - Hosp. Braga, Braga
  - Uls Regiao Leiria - Hosp. Santo Andre, Leiria
  - Uls Lisboa Ocidental - Hosp. Egas Moniz, Lisbon
  - Fund. Champalimaud, Lisbon
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Uls Loures Odivelas - Hosp. Loures, Loures
  - Hosp. Divino Espirito Santo Ponta Delgada, Ponta Delgada
  - Hosp. Cuf Porto, Porto
  - Hosp. Central Trofa Saude, Touguinho
- Romania (8):
  - Spitalul Clinic de Psihiatrie Prof Dr Alexandru Obregia, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Centrul Medical Melchisedec, Craiova
  - CMI Dr. Sarpe Marcel-Claudiu, Focşani
  - Institutului Regional de Psihiatrie 'Socola' Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Oradea, Oradea
  - Spitalul de Psihiatrie si Neurologie Brasov, Sânpetru
  - Spitalul Clinic De Psihiatrie Doctor Gheorghe Preda, Sibiu
- Serbia (5):
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Hospital Center Dr Dragisa Misovic- Dedi, Belgrade
  - Special Hospital for Psychiatric Diseases Gornja Toponica, Gornja Toponica
  - Special Hospital for Psychiatric Diseases Kovin, Kovin
  - Specialized Hospital for Psychiatric Diseases Sveti Vracevi, Novi Kneževac
- Slovakia (6):
  - Psychiatricka Ambulancia Mentum S.R.O., Bratislava
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Liptovska Nemocnica S Poliklinikou Mudr. Ivana Stodolu, Liptovský Mikuláš
  - Psychiatricka Ambulancia Psycholine S.R.O., Rimavská Sobota
  - Psychiatricka Ambulancia Centrum Zdravia R.B.K. S.R.O., Svidník
  - Crystal Comfort s.r.o., Vranov nad Topľou
- Spain (9):
  - Institucion Hosp Hestia Palau, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Gral. de Villalba, Collado Villalba
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. de Torrevieja, Torrevieja
- Sweden (4):
  - ProbarE i Lund AB, Lund
  - CTC GoCo, Mölndal
  - ProbarE i Stockholm AB, Stockholm
  - CTC MTC Uppsala, Uppsala
- Turkey (Türkiye) (10):
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Uludag Universitesi Tıp Fakultesi Hastanesi, Bursa
  - Bursa High Speciality Training and Research Dortcelik Mental Hospital, Bursa
  - Gaziantep Universitesi Tip Fakultesi, Gaziantep
  - Erenkoy Mental Hospital, Istanbul
  - Kocaeli University Medical Faculty, Kocaeli
  - Liv Hospital, Samsun
  - Karadeniz Teknik University Medical Faculty, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www janssen, com/clinical-trialsitransparency. As noted on this site, requests for access to the study data can be submitted through 'Yale Open Data Access (YODA) Project site at yoda yale.edu
URL: https://www.janssen.com/clinical-trials/transparency